CLINICAL TRIAL: NCT03556800
Title: A Phase I, Randomized, Open-Label, Single Center, Cross-over Study to Investigate the Pharmacokinetics and Safety Following a Single Application of Three Different Doses 0.5 gm (0.5 mg Estradiol), 0.75 gm (0.75 mg Estradiol) and 1.25 gm (1.25 mg Estradiol), a Transdermal Estradiol Cream (VML-0203), in Comparison to a Single Dose of EstroGelTM 1.25 gm (1 Unit/0.75 mg of Estradiol) to Healthy Post-menopausal Women.
Brief Title: Study to Investigate the Pharmacokinetics & Safety Following One Application of 3 Different Doses 0.5,0.75,& 1.25 gm,a Transdermal Estradiol Cream (VML-0203), in Comparison to a Single Dose of EstroGel 1.25 gm to Healthy Post-menopausal Women.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Viramal Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: VML-0203-002
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Menopause
Keywords: Hypoestrogenism; Menopausal hormone therapy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.5 gm of EstroCream (VML-0203) (Experimental)
  Interventions: Drug: Estrogel
- 0.75 gm of EstroCream (VML-0203) (Experimental)
  Interventions: Drug: Estrogel
- 1.25 gm of EstroCream (VML-0203) (Experimental)
  Interventions: Drug: Estrogel
- 1.25 EstroGel (Active Comparator)
  Interventions: Drug: Estrogel

INTERVENTIONS:
Drug: Estrogel — Each subject will receive the following IMPs in accordance with the randomisation code:
  * Test IMP: a single-dose of 0.5g, 0.75g and 1.25g VML-0203 cream
  * Reference IMP: a single-dose of 1.25g EstroGel
  Other Names: EstroCream

SUMMARY:
This study is a Phase I, Randomized, Open-Label, Single Center, Cross-over Study to Investigate the Pharmacokinetics and Safety following a Single Application of Three Different Doses 0.5 gm (0.5 mg estradiol), 0.75 gm (0.75 mg estradiol) and 1.25 gm (1.25 mg estradiol), a Transdermal Estradiol Cream (VML-0203), in comparison to a single dose of EstroGelTM 1.25 gm (1 unit/0.75 mg of estradiol) to healthy post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal (surgical or natural) female defined as:
* No menstrual period within the past year before study entry.
* Serum estradiol levels between 0-20 pg/ml.
* FSH levels greater than 25.8 mIU/ml.
* Greater than 45 years of age or if surgical menopausal, > 30 yrs. of age.
* Have a body mass index (BMI) between 18 and 30 kg/m2. Have had a normal PAP smear test result in line with the following guidelines:

  * aged 30 to 49 - within the last 3 years
  * aged 50 to 65 - within the last 5 years

Exclusion Criteria:

* Is pregnant (urine pregnancy test at screening) or lactating.
* Has evidence of drug or alcohol abuse.
* Have used hormonal replacement or vaginal hormonal therapy within the past three months before study entry.
* Have used estrogen pellet therapy or progestin injectable drug therapy within the past three months before study entry.
* Has contraindications to HRT use, including: unexplained vaginal bleeding, liver disease, breast or endometrial cancer, venous thromboembolic events.
* Any subjects with an obvious presence of skin conditions, excessive hair at the application sites (no shaving), scar tissue, tattoo, or coloration that would interfere with application of IMP, skin assessment, or reactions to drug.
* Presence of open sores at the application sites.
* Any subjects with a history of significant skin disorder.
* Smoker.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the bio-availability of estradiol and estrone. | 4 weeks
  Blood samples will be analysed.

SECONDARY OUTCOMES:
To provide general safety information for VML-0203. | 4 weeks
  Application site inspections will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Simona Fiore, MD, Study Director — Sponsor GmbH
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided